CLINICAL TRIAL: NCT03425513
Title: Hepatitis B Virus Prevalence and Risk Factors in Middle Limburg Belgium: the Importance of Migration.
Brief Title: Hepatitis B Virus Prevalence and Risk Factors in Belgium
Acronym: HBVBE
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Clinical Associate Professor, Hasselt University
Other Study IDs: HBVBE
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B
Keywords: Belgium; Prevalence; Risk factor; Ethnicity; Linkage of care
MeSH Terms: conditions — Hepatitis B | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatitis B group
  Interventions: Diagnostic Test: Hepatitis B serology; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Hepatitis B serology — A serum specimen will be taken and assessed for hepatitis B serology (HBsAg and anti-HBc antibodies).
Other: Questionnaire — Participants will be asked to fill in a questionnaire regarding demographic characteristics, known viral hepatitis status and risk factors for HBV infection.

SUMMARY:
The aim of this study was to evaluate the current prevalence and risk factors of hepatitis B virus (HBV) infection in a multi-ethnic neighbourhood situated in Middle Limburg, Belgium. Additionally, the investigators will determine linkage of care in hepatitis B surface antigen (HBsAg) positive subjects.

DETAILED DESCRIPTION:
Although the HBV prevalence is generally low in Western countries, such as Belgium, pockets of higher HBV prevalence exist in areas with large immigrant populations. Therefore national prevalence figures can underestimate the burden of HBV infection. The prevalence of chronic HBV in the population-based study in 2003 is believed to be an underestimate due to under-representation of the non-Belgian population. Moreover, by this time there are no data regarding the risk factors for HBV infection in the general population of Belgium.

Even in low-prevalence areas such as Belgium, HBV prevention and control is a public health priority, particularly since safe and effective vaccines are available. The aim of this study was to evaluate the current prevalence and risk factors of HBV infection in a multi-ethnic neighbourhood situated in Middle Limburg, Belgium. Additionally, the investigators will determine linkage of care in hepatitis B surface antigen (HBsAg) positive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Males and females

Exclusion Criteria:

/

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients between the age of 18 and 70 who presented at the emergency department of Ziekenhuis Oost-Limburg, a large hospital in Genk, situated in Middle Limburg.
Sampling Method: Probability Sample
Enrollment: 1131 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of current HBV infection in the Middle Limburg population | 1 day
  Serum HBsAg
Seroprevalence of past or current HBV infection in the Middle Limburg population | 1 day
  Serum anti-HBc antibodies

SECONDARY OUTCOMES:
Assess risk factors for current HBV infection in the Middle Limburg population | 1 day
  Combine results from (1) serum HBsAg with (2) questionnaire regarding demographic characteristics, known viral hepatitis status and risk factors for HBV infection.
Assess risk factors for past or current HBV infection in the Middle Limburg population | 1 day
  Combine results from (1) serum anti-HBc antibodies with (2) questionnaire regarding demographic characteristics, known viral hepatitis status and risk factors for HBV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, M.D., Ph.D., Principal Investigator — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided